CLINICAL TRIAL: NCT00003073
Title: A Phase I Dose Escalation Study of Intrathecal DepoFoam Encapsulated Cytarabine (DTC 101) in Pediatric Patients With Advanced Meningeal Malignancies
Brief Title: Chemotherapy in Treating Young Patients With Recurrent or Refractory Meningeal Leukemia, Lymphoma, or Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065754; SKYEPHARMA-96-002; DTC-96-002; NCI-V97-1336
Record Dates: First submitted 1999-11-01; First posted 2004-02-06 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2002-04

CONDITIONS: Brain and Central Nervous System Tumors; Leukemia; Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; unspecified childhood solid tumor, protocol specific; recurrent/refractory childhood Hodgkin lymphoma; leptomeningeal metastases; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Recurrence; Meningeal Carcinomatosis; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating

INTERVENTIONS:
Drug: liposomal cytarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of liposomal cytarabine in treating young patients who have recurrent or refractory meningeal leukemia, lymphoma, or solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the qualitative or quantitative toxic effects and tolerability of liposomal cytarabine (Depofoam encapsulated cytarabine; DTC 101) in pediatric patients with recurrent or refractory meningeal malignancies. II. Define a safe dose of DTC 101 in these patients for future clinical studies. III. Determine the plasma and CSF pharmacokinetics of DTC 101 in these patients.

OUTLINE: This is a dose escalation, multicenter study. Patients are placed in one of three age-related strata: stratum 1, 3 to 21 years of age; stratum 2, at least 2 but less than 3 years of age; stratum 3, at least 1 but less than 2 years of age. Patients receive an induction dose of intrathecal liposomal cytarabine (Depofoam encapsulated cytarabine; DTC 101) administered once every 2 weeks for 2 courses. Patients who have achieved a partial response or received significant clinical benefit with stable disease may receive a third induction dose of DTC 101, 2 weeks following the second dose. In the absence of progressive disease, patients can proceed to consolidation therapy. During consolidation therapy, intrathecal DTC 101 is administered once every 4 weeks for 2 courses, beginning 4 weeks after the last induction dose. Patients experiencing a complete or significant response can proceed to maintenance therapy. Patients receive a maintenance dose of intrathecal DTC 101 once every 8 weeks for a total of 6 doses, beginning 4 weeks after the second consolidation dose. At least 3 patients are evaluated at each dose level. Dose escalation to the next level proceeds when a minimum of 3 patients per cohort has successfully completed induction therapy and been evaluated. Patients will be followed at 1, 2, 3, 6, 9, and 12 months post treatment, until relapse or death.

PROJECTED ACCRUAL: A minimum of 12-15 patients will be accrued for each stratum over 18 to 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory leukemia, lymphoma, or other solid tumor that has overt meningeal involvement Definition of meningeal disease: Leukemia/lymphoma: CSF cell count at least 5/mm3 and evidence of blast cells on cytospin preparation or cytology Solid tumors: Presence of tumor cells on cytospin preparation or cytology OR evidence of meningeal disease on CT or MRI scan No bone marrow disease

PATIENT CHARACTERISTICS: Age: 1 to 21 Performance Status: ECOG 0-2 Life Expectancy: At least 8 weeks Hematopoietic: Platelet count greater than 40,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL ALT less than 5 times upper limit of normal Renal: Creatinine less than 1.5 mg/dL Other: Not pregnant or nursing Negative pregnancy test Effective contraceptive method used by fertile patients No uncontrolled illness or infection (except for HIV positive patients) No obstructive hydrocephalus or compartmentalization of the CSF flow

PRIOR CONCURRENT THERAPY: Biologic therapy: No acute toxic effects from prior immunotherapy No prior allogeneic or autologous bone marrow transplantations within 3 months of study Chemotherapy: No prior systemic CNS directed chemotherapy within 3 weeks of study No prior nitrosourea within 6 weeks of study No prior intrathecal chemotherapy within 1 week of study No acute toxic effects from prior chemotherapy No prior DTC 101 Concurrent systemic chemotherapy for management of primary cancer allowed Concurrent dexamethasone with systemic chemotherapy regimen allowed No concurrent chemotherapy for leptomeningeal disease No concurrent high dose methotrexate, high dose cytarabine, mercaptopurine, thiotepa, fluorouracil, and topotecan Endocrine therapy: Concurrent prednisone therapy with systemic chemotherapy allowed Radiotherapy: No prior craniospinal irradiation within 8 weeks of study No acute toxic effects from prior radiotherapy Concurrent local radiation therapy allowed No concurrent whole brain or craniospinal radiotherapy Surgery: Not specified Other: At least 2 weeks since investigational drugs and recovered No other concurrent investigational drugs Concurrent antibiotic therapy allowed

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 1997-02

CONTACTS AND LOCATIONS:
Overall Officials: John E. Gait, MD, Study Chair — Pacira Pharmaceuticals, Inc
Locations (6):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Alberta Children's Hospital, Calgary, Alberta, Canada